CLINICAL TRIAL: NCT05641805
Title: An Investigation of the Relationship Between Physical Activity Level and Cognitive Functions in Children With Duchenne Muscular Dystrophy
Brief Title: Physical Activity Level and Cognitive Functions in Children With Duchenne Muscular Dystrophy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Muş Alparslan University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor
Other Study IDs: GO-22/1011
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: muscular dystrophy; physical activity; cognitive function
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Motor Activity | interventions — Mental Status and Dementia Tests; Body Mass Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duchenne Muscular Dystrophy
  Interventions: Other: PAQ-C (Physical activitiy questionare for children), MoCA (Montreal Cognitive Assessment), PBS (Pediatric Balance Scale), Modified Mini Mental State Examination, BMI (Body Mass Index)

INTERVENTIONS:
Other: PAQ-C (Physical activitiy questionare for children), MoCA (Montreal Cognitive Assessment), PBS (Pediatric Balance Scale), Modified Mini Mental State Examination, BMI (Body Mass Index) — PAQ-C will use to evaluate physical activity level of participants. MoCA and Modified Mini Mental State Examination will use to evaluate cognitive functions of participants.
  PBS will use to evaluate participants' balance responses.

SUMMARY:
Although there are studies showing that the effect on motor performance over time in children with DMD is associated with a decrease in the level of physical activity, no publication has been found that directly examines the relationship between cognitive functions and physical activity level. Therefore, the aim of our study is to investigate the relationship between physical activity level and cognitive functions in children with DMD.

DETAILED DESCRIPTION:
In DMD; as a result of mutations in the Xp21.2 region of the dystrophin gene, which encodes the dystrophin protein, which plays an important role in the normal contraction and relaxation of the muscle, progressive weakness starting from the proximal extremity muscles, chronic degeneration, replacement of the muscle with fat and connective tissue occurs due to the production of deficient or fully functional dystrophin. Although motor performance is one of the most prominent features in children with DMD, it has been reported that cognitive functions are also significantly affected in one third of children compared to their healthy peers. In addition, the physical activity levels of children with DMD show a significant decrease in physical activity levels after the age of 5, when motor problems are more pronounced than their healthy peers. Recently, interest in studies on physical activity level and cognitive skills in pediatric neuromuscular diseases such as DMD has increased, and studies have revealed the relationship between cognitive functions and motor performance. There are also studies showing that the effect on motor performance over time is associated with a decrease in physical activity level. However, there are no publications that directly examine the relationship between cognitive functions and physical activity level in children with DMD. Therefore, the primary aim of our study is; to investigate the relationship between physical activity level and cognitive functions in children with DMD. The secondary aims of our study are to reveal the relationship between balance and body mass index and physical activity level in children with DMD.

ELIGIBILITY:
Inclusion Criteria:

* Children who diagnosed with Duchenne Muscular Dystrophy (DMD), between the ages of 8-14, to have cognitive functions at a level to understand and apply test directives, Level 1-5 according to Brooke lower extremity functional classification will be included.

Exclusion Criteria:

* Children who have any chronic or systemic disease in addition to DMD, being above level 5 according to the Brooke lower extremity functional classification, have a cooperation problem, have had any lower/upper extremity injury and/or surgery in the last 6 months and children who did not give consent will be excluded.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Ambulatory children with Duchenne muscular dystrophy, between the ages of 8-14
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
PAQ-C | 10 to 15 minutes
  Physical activity level
MoCA | 10 to 15 minutes
  Cognitive function
Modified Mini Mental State Examination | 10 to 15 minutes
  Cognitive function

SECONDARY OUTCOMES:
PBS | 10 to 15 minutes
  Balance responses of participants
BMI | 1 minute
  Body mass index to evaluate weight status of participants

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Sırrı, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided